CLINICAL TRIAL: NCT05299424
Title: A Multi-center, Open-label, Phase 1/2 Clinical Study of CM336 Injection in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of CM336 in Patients With Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CM336-021001
Record Dates: First submitted 2022-02-17; First posted 2022-03-29 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1, Dose escalation (Experimental): There are 14 dose groups in dose escalation part ( Phase 1 study).
  Interventions: Drug: CM336_group 1; Drug: CM336_group 2a; Drug: CM336_group 2b; Drug: CM336_group 3a; Drug: CM336_group 3b; Drug: CM336_group 4a; Drug: CM336_group 4b; Drug: CM336_group 5; Drug: CM336_group 6a; Drug: CM336_group 6b; Drug: CM336_group 7; Drug: CM336_group 8a; Drug: CM336_group 8b; Drug: CM336_group 9
- Phase 2, Dose expansion (Experimental): Based on the data of phase 1, the dose level recommended for the phase 2 study (RP2D) will be evaluated.
  Interventions: Drug: CM336_RP2D

INTERVENTIONS:
Drug: CM336_group 1 — CM336 will be administered subcutaneously (SC) once a week (QW). Patients will take 0.04mg of CM336 on the first day of first cycle (C1D1), 0.04mg on C1D8, 0.04mg on C1D15 and subsequent treatment cycles until there is evidence of disease progression, unacceptable toxicity or other reasons for treatment discontinuation.
  Arms: Phase 1, Dose escalation
Drug: CM336_group 2a — CM336 will be administered subcutaneously (SC) once a week (QW). Patients will take 0.04mg of CM336 on the first day of first cycle (C1D1), 0.2mg on C1D8, 1.0mg on C1D15 and subsequent treatment cycles until there is evidence of disease progression, unacceptable toxicity or other reasons for treatment discontinuation.
  Arms: Phase 1, Dose escalation
Drug: CM336_group 2b — CM336 will be administered subcutaneously (SC) once a week (QW). Patients will take 0.2mg of CM336 on the first day of first cycle (C1D1), 0.2mg on C1D8, 0.2mg on C1D15 and subsequent treatment cycles until there is evidence of disease progression, unacceptable toxicity or other reasons for treatment discontinuation.
  Arms: Phase 1, Dose escalation
Drug: CM336_group 3a — CM336 will be administered subcutaneously (SC) once a week (QW). Patients will take 0.2mg of CM336 on the first day of first cycle (C1D1), 1.0mg on C1D8, 5.0mg on C1D15 and subsequent treatment cycles until there is evidence of disease progression, unacceptable toxicity or other reasons for treatment discontinuation.
  Arms: Phase 1, Dose escalation
Drug: CM336_group 3b — CM336 will be administered subcutaneously (SC) once a week (QW). Patients will take 1.0mg of CM336 on the first day of first cycle (C1D1), 1.0mg on C1D8, 1.0mg on C1D15 and subsequent treatment cycles until there is evidence of disease progression, unacceptable toxicity or other reasons for treatment discontinuation.
  Arms: Phase 1, Dose escalation
Drug: CM336_group 4a — CM336 will be administered subcutaneously (SC) once a week (QW). Patients will take 1.0mg of CM336 on the first day of first cycle (C1D1), 5.0mg on C1D8, 15.0mg on C1D15 and subsequent treatment cycles until there is evidence of disease progression, unacceptable toxicity or other reasons for treatment discontinuation.
  Arms: Phase 1, Dose escalation
Drug: CM336_group 4b — CM336 will be administered subcutaneously (SC) once a week (QW). Patients will take 2.0mg of CM336 on the first day of first cycle (C1D1), 2.0mg on C1D8, 2.0mg on C1D15 and subsequent treatment cycles until there is evidence of disease progression, unacceptable toxicity or other reasons for treatment discontinuation.
  Arms: Phase 1, Dose escalation
Drug: CM336_group 5 — CM336 will be administered subcutaneously (SC) once a week (QW). Patients will take 2.0mg of CM336 on the first day of first cycle (C1D1), 8.0mg on C1D8, 24.0mg on C1D15 and subsequent treatment cycles until there is evidence of disease progression, unacceptable toxicity or other reasons for treatment discontinuation.
  Arms: Phase 1, Dose escalation
Drug: CM336_group 6a — CM336 will be administered subcutaneously (SC) once a week (QW). Patients will take 2.0mg of CM336 on the first day of first cycle (C1D1), 10.0mg on C1D8, 40.0mg on C1D15 and subsequent treatment cycles until there is evidence of disease progression, unacceptable toxicity or other reasons for treatment discontinuation.
  Arms: Phase 1, Dose escalation
Drug: CM336_group 6b — CM336 will be administered subcutaneously (SC) once a week (QW). Patients will take 3.0mg of CM336 on the first day of first cycle (C1D1), 3.0mg on C1D8, 3.0mg on C1D15 and subsequent treatment cycles until there is evidence of disease progression, unacceptable toxicity or other reasons for treatment discontinuation.
  Arms: Phase 1, Dose escalation
Drug: CM336_group 7 — CM336 will be administered subcutaneously (SC) once a week (QW). Patients will take 3.0mg of CM336 on the first day of first cycle (C1D1), 15.0mg on C1D8, 60.0mg on C1D15 and subsequent treatment cycles until there is evidence of disease progression, unacceptable toxicity or other reasons for treatment discontinuation.
  Arms: Phase 1, Dose escalation
Drug: CM336_group 8a — CM336 will be administered subcutaneously (SC) once a week (QW). Patients will take 3.0mg of CM336 on the first day of first cycle (C1D1), 15.0mg on C1D8, 75.0mg on C1D15 and subsequent treatment cycles until there is evidence of disease progression, unacceptable toxicity or other reasons for treatment discontinuation.
  Arms: Phase 1, Dose escalation
Drug: CM336_group 8b — CM336 will be administered subcutaneously (SC) once a week (QW). Patients will take 4.0mg of CM336 on the first day of first cycle (C1D1), 4.0mg on C1D8, 4.0mg on C1D15 and subsequent treatment cycles until there is evidence of disease progression, unacceptable toxicity or other reasons for treatment discontinuation.
  Arms: Phase 1, Dose escalation
Drug: CM336_group 9 — CM336 will be administered subcutaneously (SC) once a week (QW). Patients will take 4.0mg of CM336 on the first day of first cycle (C1D1), 20.0mg on C1D8, 90.0mg on C1D15 and subsequent treatment cycles until there is evidence of disease progression, unacceptable toxicity or other reasons for treatment discontinuation.
  Arms: Phase 1, Dose escalation
Drug: CM336_RP2D — CM336 will be administered subcutaneously (SC) once a week (QW). Individual subjects may continue study treatment until disease progression/relapse, unacceptable toxicity, withdrawal of consent, receipt of other anti-MM therapies, death, loss to follow-up, or the end of study.
  Arms: Phase 2, Dose expansion

SUMMARY:
This is a multi-center, open-label, Phase 1/2 study in China to evaluate the safety, tolerability, efficacy, pharmacokinetics, pharmacodynamics and immunogenicity of CM336 in patients with relapsed or refractory multiple myeloma.

This study consists of a dose escalation part (Phase 1) and a dose extension part (Phase 2 ).

The safety and tolerability of CM336 will be evaluated in Phase 1 study, as well as the maximum tolerated dose (MTD) and the recommended dose level for Phase 2 study will be determined.

The efficacy of CM336 will be evaluated in Phase 2 study.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group Performance Status (ECOG) of 0-2.
* Patients with relapsed or refractory MM who have failed or are intolerant to all therapies with known clinical benefit; patients must have received at least 2 prior anti-myeloma therapies which must contain at least one proteasome inhibitor (PI), one immunomodulatory drug (IMiD), and one anti-CD38 monoclonal antibody (if available).

Exclusion Criteria:

* Patients who had received BCMA-targeted therapy.
* Patients who had received CAR-T therapy.
* Patients who had received anti-tumor therapy within 3 weeks or 5 half-lives (whichever is shorter) prior to the first dose of CM336.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-08-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) | 21 days after the first dose
  Dose-limiting toxicities (DLTs)
Adverse events (AEs) | Up to 4.5 years
  Adverse events (AEs), including any abnormal physical examinations, abnormal vital signs, abnormal ECG, and abnormal lab testing.
Overall Response Rate (ORR) | up to 4.5 years
  Assessed according to International Myeloma Working Group (IMWG) response criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Hongmei Jing, Principal Investigator — Peking University Third Hospital; Lugui Lugui, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China